CLINICAL TRIAL: NCT06438146
Title: Liraglutide for Management of Obesity in People Living With HIV on Dolutegravir-based Antiretroviral Therapy: a Single-arm Acceptability Study in South Africa
Brief Title: LIROH - Liraglutide for Obesity in HIV
Acronym: LIROH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer M. Manne-Goehler, MD, SCD, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002985; K23DK125162 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Obesity; HIV Infections
Keywords: HIV; Obesity; Liraglutide; Behavior; Exercise; Lifestyle counseling
MeSH Terms: conditions — Obesity; HIV Infections; Behavior; Motor Activity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lirgalutide (Experimental): Following individual informed consent, all participants will undergo a series of basic cardiometabolic labs. They will then be initiated on liraglutide 0.6 mg administered subcutaneously, and this dose will be gradually increased over a period of 4 weeks to a dose of 3.0mg daily. Alongside drug administration, participants will receive lifestyle counselling regarding diet and physical activity. Following completion of a 12-week "on treatment" period, liraglutide will be stopped and participants will be followed for an additional 12-weeks off treatment. Body weight, cardiometabolic risk parameters, and a suite of patient-reported outcomes regarding diet, physical activity, sleep, and quality of life will be assessed periodically over the course of the study.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Dosing regimen: In this study protocol, liraglutide dosing will be implemented as follows: Liraglutide will be started at a dose of 0.6 mg per day. Participants will be taught to use the injection pen and will be observed giving the first injection. The dose will then be increased by 0.6 mg each week to a maximum dosage of 3.0 mg per day at the end of 4 weeks.
  This corresponds to the following dosing schedule:
  Week 1: 0.6 mg per day for one week Week 2: 1.2 mg per day for one week Week 3: 1.8 mg per day for one week Week 4: 2.4 mg per day for one week Week 5-12: 3.0 mg per day for 8 weeks Week 13-24: No drug administration
  Other Names: Saxenda

SUMMARY:
The goal of this single-arm, open label pilot study is to evaluate liraglutide at the recommended dosage administered subcutaneously + lifestyle counselling for the management of people living with HIV (PLWH) with obesity defined by a BMI ≥30 kg/m2 who are on dolutegravir-based ART.

Following individual informed consent, all participants will undergo a series of basic cardiometabolic labs. They will then be initiated on liraglutide 0.6 mg administered subcutaneously, and this dose will be gradually increased over a period of 4 weeks to a dose of 3.0 mg daily. Alongside drug administration, participants will receive lifestyle counselling regarding diet and physical activity. Following completion of a 12-week "on treatment" period, liraglutide will be stopped and participants will be followed for an additional 12-weeks off treatment. Body weight, cardiometabolic risk parameters, and a suite of patient-reported outcomes regarding diet, physical activity, sleep, and quality of life will be assessed periodically over the course of the study.

DETAILED DESCRIPTION:
South Africa has the largest population of PLWH globally, with a prevalence of 17% in adults or 7.2 million PLWH. The rapid scale-up of ART programs has resulted in >6 million PLWH on treatment, significant gains in life expectancy, and a large population of aging PLWH. With increasing life expectancy, obesity and type 2 diabetes have become growing threats for PLWH in South Africa and globally. One recent study found that 63% of PLWH are overweight or obese, and 6% have diabetes in this setting.

This elevated risk of obesity in PLWH in South Africa is likely due to a confluence of both general considerations and HIV-specific factors. First, South Africa has experienced an accelerated background epidemic of metabolic disease in the general population with a prevalence of overweight and obesity that is nearly equal to that of high-income countries. Additionally, the International Diabetes Federation estimates that approximately 15.5 million adults are living with diabetes in the African Region, and projects it to grow to 41 million by 2045. As part of this background epidemic of metabolic disease, South Africa is also experiencing a nutrition transition, with widespread availability of processed and refined foods as well as sugar-sweetened beverages.

Regarding HIV-specific issues, in 2019 the first-line ART regimen for the South African national HIV treatment program transitioned to TLD. TLD is generally very safe and well-tolerated and has a high barrier to HIV resistance but this transition to this regimen has been associated with risk of excess weight gain at the population level. Both clinical trials and observational studies conducted in South Africa have shown substantial increases in body weight in those who are initiating this ART regimen newly and among those who are suppressed and switched, especially women. Given this, there is a growing risk of obesity in PLWH in this context and a need for management strategies to address this increasingly prevalent comorbidity.

Preventing the metabolic complications of HIV in South Africa and worldwide requires urgent solutions. To date, obesity management and diabetes prevention have largely consisted of behavioural interventions such as the Diabetes Prevention Program and related lifestyle modification efforts, focused on improving diet and increasing physical activity. However, in the past several years, novel anti-obesity pharmacologic agents such as the glucagon-like peptide-1 receptor agonists (GLP-1 RAs) have shown enormous promise for obesity management and diabetes prevention in people who are HIV-negative (8-10). However, this drug class has a very limited evidence base in PLWH and relatively scant data from sub-Saharan African populations.

Currently, liraglutide is the only GLP-1 RA approved for obesity management in South Africa and this protocol proposes to use the drug for its labelled indication of "weight loss in addition to diet and exercise in adults aged 18 and above who have: (1) a BMI of 30 or greater (obese) or (2) a BMI of greater than 27 and less than 30 (overweight) and weight related health problems (such as diabetes, high blood pressure, hypercholesterolemia, or obstructive sleep apnoea).

This evidence gap motivates further inquiry into GLP-1 RAs such as liraglutide as one potential approach to obesity management and prevention of diabetes in PLWH who have comorbid obesity in South Africa, with implications for PLWH in other contexts. In this proposal, the investigators seek to further this important area of inquiry by evaluating the acceptability of liraglutide along with lifestyle counselling in PLWH who have obesity and are stable on dolutegravir-based ART in South Africa.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent to participate in the study
2. Able to comply with all study procedures, including daily subcutaneous injections
3. Adults ≥18 years old
4. PLWH on dolutegravir-based ART for ≥6 months
5. Documented HIV-1 viral load in the past 6 months confirming the participant is virologically suppressed
6. BMI ≥30 kg/m2
7. Desiring weight loss
8. Willing to undertake lifestyle change
9. Not on any weight loss agent for the duration of the study

Exclusion Criteria:

1. Self-reported history of diabetes
2. Current use of medications for diabetes
3. Known contraindications to liraglutide, such as hypersensitivity to a component of the drug
4. Current pregnancy or desire to become pregnant
5. History of pancreatitis
6. History of thyroid disease
7. History of harmful use of alcohol
8. Clinically unstable in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who screen and enroll among those approached | Measured at screening
  This will be expressed in terms of the proportion of participants who attend screening and enrolment visits among the total number who are approached regarding interest in study participation.
Time to reach study enrollment target | Measured at enrollment
Study retention rate at 12 weeks | Measured at Visit 4 at 12 weeks
  This will be expressed as a proportion of participants who remain in the study after the 12 week "on treatment" period among those enrolled.
Study retention rate at 24 weeks | Measured at End of Study at 24 weeks
  This will be expressed as a proportion of participants who remain in the study after the full 24 weeks of study procedures are completed among those enrolled.
Rate of adherence to treatment over 12 weeks | Measured at Visit 4 at 12 weeks
  The investigators will assess volume remaining in the injector pens and provide a percentage of doses per participant that remained unused at the end of the 12-week period on treatment.
Embedded qualitative interviews regarding the acceptability of liraglutide for obesity management | Measured at End of Study at 24 weeks
  This will be open-ended responses to a brief exit interview about acceptability and feasibility.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events as defined in this protocol | From the initiation of treatment until the date of a treatment-emergent adverse event, assessed up to 24 weeks.
  The investigators will report incidence of TEAEs up to 24 weeks (12 weeks on + 12 weeks off treatment)
Incidence of serious adverse events (SAEs), as defined in this protocol | From the initiation of treatment until the date of a serious adverse event, assessed up to 24 weeks.
  The investigators will report incidence of SAEs up to 24 weeks (12 weeks on + 12 weeks off treatment)
Change in body weight following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  Body weight will be measured in the study at both enrolment and after 12 weeks on treatment (Visit 4); these will be used to calculate a continuous change in kg.
Change in body weight over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  Body weight will be measured in the study at both enrolment and after 24 weeks on treatment (EOS); these will be used to calculate a continuous change in kg.
Change in HbA1c following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  HbA1c will be measured at enrolment and at Visit 4; here investigators will calculate the difference between these measures (in %).
Change in HbA1c over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  HbA1c will be measured at enrolment and at EOS; here investigators will calculate the difference between these measures (in %).
Change in fasting plasma glucose following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  Fasting glucose will be measured at enrolment and at Visit 4; investigators will calculate the difference between these measures (in mmol/L).
Change in fasting plasma glucose over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  Fasting glucose will be measured at enrolment and at EOS; investigators will calculate the difference between these measures (in mmol/L).
Change in depressive symptoms following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  This will be defined as the difference in depression score per the Patient Health Questionnaire (PHQ-9) at enrolment and Visit 4. The minimum value is 1 and the maximum is 27, where the greater the total score, the greater severity of depression.
Change in depressive symptoms over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  This will be defined as the difference in depression score per the Patient Health Questionnaire (PHQ-9) at enrolment and EOS. The minimum value is 1 and the maximum is 27, where the greater the total score, the greater severity of depression.
Change in physical activity level following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  This will be defined as the difference in physical activity expressed in MET-minutes per week, where MET minutes represent the amount of energy expended carrying out physical activity, per the International Physical Activity Questionnaire (IPAQ) at enrolment and Visit 4.
Change in physical activity level over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  This will be defined as the difference in physical activity expressed in MET-minutes, where MET minutes represent the amount of energy expended carrying out physical activity, per week per the International Physical Activity Questionnaire (IPAQ) at enrolment and EOS.
Change in dietary habits following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  This will be defined as the difference in total servings of fruits and vegetables, change in frequency of sugar-sweetened beverage intake, and change frequency of fast food intake from enrolment to Visit 4.
Change in dietary habits over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  This will be defined as the difference in total servings of fruits and vegetables, change in frequency of sugar-sweetened beverage intake, and change frequency of fast food intake from enrolment to EOS.

OTHER OUTCOMES:
Change in blood pressure following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  Systolic blood pressure change in mm Hg
Change in blood pressure over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  Blood pressure change in mm Hg
Change in lipids following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  Change in total cholesterol
Change in lipids over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  Change in total cholesterol
Change in waist circumference following 12 weeks on treatment | Measured at Visit 4 at 12 weeks
  Change in waist circumference in cm
Change in waist circumference over 24 weeks (12 weeks on + 12 weeks off treatment) | Measured at End of Study at 24 weeks
  Change in waist circumference in cm
Change in quality of life following 12 weeks on treatment per the World Health Organization's Quality of Life Instrument in HIV Infection | Measured at Visit 4 at 12 weeks
  Change in quality of life scale score (scale of 0 - 100)
Change in quality of life over 24 weeks (12 weeks on + 12 weeks off treatment) per the World Health Organization's Quality of Life Instrument in HIV Infection | Measured at End of Study at 24 weeks
  Change in quality of life scale score (scale of 0 - 100)
Change in sleep quality following 12 weeks on treatment per the Pittsburgh Sleep Quality Index | Measured at Visit 4 at 12 weeks
  Change in sleep quality scale score (global score range of 0 to 21 where score of 5 or greater indicates poor sleep)
Change in sleep quality over 24 weeks (12 weeks on + 12 weeks off treatment) per the Pittsburgh Sleep Quality Index | Measured at End of Study at 24 weeks
  Change in sleep quality scale score (global score range of 0 to 21 where score of 5 or greater indicates poor sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Manne-Goehler, MD, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Africa Health Research Institute Clinical Trials Unit, Mtubatuba, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data as allowable
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD data will be shared in accordance with AHRI Data Access Policy and Data Management Plan within two years of completion.
Access Criteria: Access to the IPD and the associated documents will require completion of the online data access application form accessible on the AHRI Data repository. AHRI bona fide data users are required to abide by the data use conditions stipulated on the application for access to the data.
URL: https://data.ahri.org/

REFERENCES:
- [Background] Venter WDF, Moorhouse M, Sokhela S, Fairlie L, Mashabane N, Masenya M, Serenata C, Akpomiemie G, Qavi A, Chandiwana N, Norris S, Chersich M, Clayden P, Abrams E, Arulappan N, Vos A, McCann K, Simmons B, Hill A. Dolutegravir plus Two Different Prodrugs of Tenofovir to Treat HIV. N Engl J Med. 2019 Aug 29;381(9):803-815. doi: 10.1056/NEJMoa1902824. Epub 2019 Jul 24. PMID 31339677
- [Background] Venter WDF, Sokhela S, Simmons B, Moorhouse M, Fairlie L, Mashabane N, Serenata C, Akpomiemie G, Masenya M, Qavi A, Chandiwana N, McCann K, Norris S, Chersich M, Maartens G, Lalla-Edward S, Vos A, Clayden P, Abrams E, Arulappan N, Hill A. Dolutegravir with emtricitabine and tenofovir alafenamide or tenofovir disoproxil fumarate versus efavirenz, emtricitabine, and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection (ADVANCE): week 96 results from a randomised, phase 3, non-inferiority trial. Lancet HIV. 2020 Oct;7(10):e666-e676. doi: 10.1016/S2352-3018(20)30241-1. PMID 33010240
- [Background] Manne-Goehler J, Rahim N, van Empel E, de Vlieg R, Chamberlin G, Ihama A, Castle A, Mabweazara S, Venter WDF, Chandiwana N, Levitt NS, Siedner M. Perceptions of Health, Body Size, and Nutritional Risk Factors for Obesity in People with HIV in South Africa. AIDS Behav. 2024 Jan;28(1):367-375. doi: 10.1007/s10461-023-04152-7. Epub 2023 Aug 26. PMID 37632604
- [Background] Chandiwana NC, Siedner MJ, Marconi VC, Hill A, Ali MK, Batterham RL, Venter WDF. Weight Gain After HIV Therapy Initiation: Pathophysiology and Implications. J Clin Endocrinol Metab. 2024 Jan 18;109(2):e478-e487. doi: 10.1210/clinem/dgad411. PMID 37437159
- [Background] Magodoro IM, Olivier S, Gareta D, Koole O, Modise TH, Gunda R, Herbst K, Pillay D, Wong EB, Siedner MJ. Linkage to HIV care and hypertension and diabetes control in rural South Africa: Results from the population-based Vukuzazi Study. PLOS Glob Public Health. 2022 Nov 2;2(11):e0001221. doi: 10.1371/journal.pgph.0001221. eCollection 2022. PMID 36962629
- [Background] Rubino DM, Greenway FL, Khalid U, O'Neil PM, Rosenstock J, Sorrig R, Wadden TA, Wizert A, Garvey WT; STEP 8 Investigators. Effect of Weekly Subcutaneous Semaglutide vs Daily Liraglutide on Body Weight in Adults With Overweight or Obesity Without Diabetes: The STEP 8 Randomized Clinical Trial. JAMA. 2022 Jan 11;327(2):138-150. doi: 10.1001/jama.2021.23619. PMID 35015037
- [Background] Wadden TA, Bailey TS, Billings LK, Davies M, Frias JP, Koroleva A, Lingvay I, O'Neil PM, Rubino DM, Skovgaard D, Wallenstein SOR, Garvey WT; STEP 3 Investigators. Effect of Subcutaneous Semaglutide vs Placebo as an Adjunct to Intensive Behavioral Therapy on Body Weight in Adults With Overweight or Obesity: The STEP 3 Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1403-1413. doi: 10.1001/jama.2021.1831. PMID 33625476
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Hyle EP, Bekker LG, Martey EB, Huang M, Xu A, Parker RA, Walensky RP, Middelkoop K. Cardiovascular risk factors among ART-experienced people with HIV in South Africa. J Int AIDS Soc. 2019 Apr;22(4):e25274. doi: 10.1002/jia2.25274. PMID 30990252
- [Background] Bailin SS, Gabriel CL, Wanjalla CN, Koethe JR. Obesity and Weight Gain in Persons with HIV. Curr HIV/AIDS Rep. 2020 Apr;17(2):138-150. doi: 10.1007/s11904-020-00483-5. PMID 32072466